CLINICAL TRIAL: NCT04241991
Title: Effects of Laser Photobiomodulation (PBM) Therapy at 808 nm on Muscle Performance in Elderly Women: a Randomized, Controlled Trial
Brief Title: Photobiomodulation (PBM) Therapy on Muscle Performance in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Andreo Fernando Aguiar, Principal Investigator, Universidade Norte do Paraná
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 2.893.464
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Lasers; Resistance Training; Muscle Strength; Aged; Performance
Keywords: Photobiomodulation; Muscle function; Elderly; Resistance exercise; Balance

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and researchers used dark laser goggles for eye protection against irradiation, and participants were blinded by a blindfold on top of safety glasses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active laser (Experimental): Each participant will receive the application of the active laser on the rectus femoris muscle during the trials 1 (acute) and 2 (chronic).
  Interventions: Radiation: Active laser
- Placebo laser (Placebo Comparator): Each participant will receive the application of the placebo laser on the rectus femoris muscle during the trials 1 (acute) and 2 (chronic).
  Interventions: Radiation: Placebo laser

INTERVENTIONS:
Radiation: Active laser — Participants will receive laser irradiation on the rectus femoris muscle of both legs immediately before the test (trial 1) and training (trial 2) sessions. A researcher blinded to the treatment conditions will apply the irradiation on eight points distributed over the muscle belly, using a gallium arsenide aluminum (Ga-As-Al) laser (λ: 808 nm) equipment. The points will placed at 25, 35, 50 and 75% of the total distance between the anterior superior iliac spine and superior border of the patella, bilaterally, with 2 cm of distance between each point.
  Other Names: Active laser therapy
  Arms: Active laser
Radiation: Placebo laser — Participants will receive placebo irradiation on the rectus femoris muscle of both legs immediately before the test (trial 1) and training (trial 2) sessions. A researcher blinded to the treatment conditions will apply the placebo irradiation on eight points distributed over the muscle belly. The points will placed at 25, 35, 50 and 75% of the total distance between the anterior superior iliac spine and superior border of the patella, bilaterally, with 2 cm of distance between each point.
  Other Names: Placebo laser therapy
  Arms: Placebo laser

SUMMARY:
The present project aims to investigate the acute and chronic effects of laser photobiomodulation (PBM) at 808 nm on muscle performance in physically active elderly women. The hypothesis of this study is that laser PBM would improve muscle strength (i.e., MVIC and 1RM) and endurance (i.e., repetitions-to-failure, blood lactate levels), functional capacity (i.e., short physical performance battery score), and rating of perceived exertion when compared with placebo laser.

DETAILED DESCRIPTION:
The purpose of this study will be to investigate the acute and chronic effects of laser PBM (λ: 808 nm) on muscle performance in physically active elderly women. For this purpose, the participants will be enrolled in two trials: Trial 1: Initially, all participants (n = 20/group) will be submitted for a 1-wk familiarization period (3 non-consecutive sessions) of functional tests (i.e., standing balance, gait speed, and chair stand tests) from short physical performance battery (SPPB), knee flexion-extension exercise (3 sets of 10-12 repetitions), maximum voluntary isometric contraction (MVIC), balance test on a force platform, and one-repetition maximum (1RM) test for knee extension exercise. Thereafter, participants will be randomized to receive 1 of 2 treatments (active or placebo laser) on two occasions (T1 and T2), separated by a 7-day washout period. During T1 and T2, participants will receive their respective treatments and then perform the muscle performance tests, separated by 10 minutes, in the following order: SPPB, MVIC, and repetitions-to-failure. After the last test, the participants will be instructed to reported the perceived exertion by OMNI scale, and a blood sample will be collected for measurement of blood lactate levels. Differences between groups will be assessed using a 2-tailed paired t-test. The significance level will be 0.05. Trial 2: participants will be randomized into two groups (n = 20/group): active laser or placebo laser. Both groups will be submitted for a 10-wk resistance training program (2 x/week) involving unilateral knee extension exercise. The following variables will be assessed from pre-to post-training: anthropometric, muscle thickness from vastus lateralis muscle using ultrasound, MVIC, 1RM, repetition-to-failure, and balance variables on a force platform. Shapiro-Wilk and Levine tests will be used to test the normality and homogeneity of the measurements, respectively. Two-way ANOVA (group x time) tests for repeated measures will be performed to assess changes over time and between groups for all dependent variables. Violation of sphericity will adjust using Greenhouse-Geser correction. The Bonferroni post-hoc test will detect specific differences between groups. When appropriate, the percentage of change (∆%) will be reported according to the following equation: ∆% = [(pre-average post average) / pre-average mean] × 100. Values will be express as mean ± standard deviation. O significance level α will be 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-80 y,
* Classified as eutrophic (i.e., body mass index ≤ 27 kg/m2), and
* Classified as physically active (i.e., performing at least 150 min/week of moderate physical activity) according to criteria of the International Physical Activity Questionnaire (IPAQ) for elderly

Exclusion Criteria:

* To be tobacco product users
* To make use of any ergogenic supplement within six months prior to the start of the study;
* To make use of any medication that could affect the ability to perform the physical tests;
* To have any physiological (e.g., cardiorespiratory and metabolic diseases, uncontrolled hypertension, or diabetes) or physical limitation (e.g., orthopedic or rheumatic diseases, muscular injury, fibromyalgia, or pain) that could affect the ability to perform the physical tests, or
* To be unable to understand the informed consent document and provide a detailed description of their lifestyle.

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in vastus lateralis thickness | Baseline and after 10 weeks
  Muscle thickness measured by ultrasonography
Change in maximal dynamic strength by 1RM | Baseline and after 10 weeks
  1RM for knee extension exercise.
Change in MVIC | Immediately after intervention (Trial 1), and baseline and after 10 weeks (Trial 2)
  MVIC using a portable fixed dynamometry (i.e., compression load cell)
Change in functional capacity | Immediately after intervention (Trial 1).
  Functional capacity measured by short physical performance battery (SPPB)
Change in balance | Baseline and after 10 weeks (Trial 2)
  Balance performance using a force platform.
Change in repetitions-to-failure | Immediately after intervention (Trial 1), and baseline and after 10 weeks (Trial 2)
  Repetitions-to-failure test on a knee extension machine.

SECONDARY OUTCOMES:
Change in lactate levels | Immediately after repetitions-to-failure test (trial 1)
  Blood samples will be collected for analyse of the lactate levels after repetitions-to-failure test
Change in perceived exertion | Immediately after repetitions-to-failure test (trial 1)
  Perceived exertion after repetitions-to-failure test using the OMNI scale

CONTACTS AND LOCATIONS:
Overall Officials: Andreo Aguiar, Dr., Principal Investigator — North University of Paraná
Locations (1):
- Universidade Norte do Paraná, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No